CLINICAL TRIAL: NCT02651233
Title: Factors That May Influence Yield and Viability of Extracted Adipose Derived Regenerative Cells' Per Gram of Fat Tissue
Brief Title: Factors That Influence Adipose Derived Regenerative Cells' Yield and Viability
Status: Completed | Type: Observational
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Katarina Andjelkov, Clinical professor, principal investigator, Clinical Centre of Serbia
Other Study IDs: CCSerbia
Record Dates: First submitted 2016-01-02; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Problem of Aging; Smoking; Physical Activity; Gender
MeSH Terms: conditions — Smoking; Motor Activity; Coitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ADRCs therapy — Patients are submitted to manual liposuction and extraction of ADRCS is done with closed system. All patients were candidates for subcutaneous transplantation of autologous cell enriched adipose tissue for different indications.

SUMMARY:
Human adipose tissue has been shown to contain a group of cells that possess extensive proliferative capacity and the ability to differentiate into multiple cell lineages. Cells isolated from the fatty portion are termed processed lipoaspirate cells that contain adipose-derived regenerative cells (ADRCs). ADRCs are most conveniently extracted from tissue during an elective cosmetic liposuction procedure but may also be obtained from resected adipose tissue.

This study is aimed to verify if there are differences between the number and viability of cells obtained from patients with different age, sex, Body Mass Index (BMI), smoking and physical activity, within the different amount of processed fat.

DETAILED DESCRIPTION:
Method: We analyzed 46 patients, both sexes, who filled out a questionnaire about their age and habits (sport activity and smoking). They were then divided into two groups. Group 1 consisted of patients with normal BMI range from 18,5 to 24.9 (n=27) and Group 2 had overweight patients with BMI index 25 to 29.9 (n=19). There were no underweight or obese patients. All 46 patients had the ADRCS extracted for therapeutical use, but with different indications. The mixture of 180 mL saline solution, 1mL Epinephrine (1:10,000) and 20 mL of 2% lidocaine is injected in the subcutaneous layer of the abdominal wall to allow the tumescence and to decrease the blood loss. The manual liposuction procedure has been carried out through two or three small incisions using harvester (Tulip® medical products, San Diego, USA). All of them had liposuction done by the author and in the same manner (tumescent technique, same cannula) to obtain 120-200ml of fat. The harvest site is then covered with a pressure dressing for 10 days to reduce swelling and hematoma. The closed system PureGraft® 250mL (PureGraft®, Solana Beach, California, USA) has been used used to collect the specimen. The specimen is transferred within 15 min to the BelPrime Clinic laboratory where the Celution® 800/CRS system (Cytori Therapeutics, Inc. San Diego, California, USA) is applied to process the lipoaspirate in order to obtain ADRCs. The Celution® 800/CRS system is a closed automated medical device that helps to separate blood and fat. The system will then digests fat using the proprietary enzyme reagent Celase 835/CRS (Cytori Therapeutics, Inc. San Diego, California, USA) to release the stromal vascular fraction (SVF). SVF is subsequently concentrated by a short centrifugation and then automated wash cycles to obtain the ADRC fraction. This 90 to 120-minute process provides approximately 5mL of pellet. A few drops of the obtained pellet were immediately used for cell counting (ChemoMetec A/S DK-3450, Allerod, Denmark).

Results/Complications: Number of ADRCS obtained, cells' viability, viable ADRCS per gram of fat processed, ADRCS for active dose and total volume for cell therapy were statistically analyzed in correlation with patients' BMI, sport activity, sex, age and smoking habits and amount of processed fat.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were: healthy individuals, both genders, there were no age nor BMI restriction, smokers and no smokers searching for local, subcutaneous transplantation of ADRCs.

Exclusion Criteria:

The exclusion criteria were autoimmune diseases, inflammatory bowel disease, presence of malignant or chronic infectious disease, or immunosuppressive therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients were healthy individuals, both genders with request for subcutaneous transplantation of autologous cell enriched adipose tissue for different indications
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (Calculated in kg/m2) | 1h before the surgery
  Calculated in kg/m2

SECONDARY OUTCOMES:
ADRCs yield (Calculated in number of cells per gram of tissue) | 2h after the surgery
  Calculated in number of cells per gram of tissue
ADRCs viability (Calculated in percentage) | 2h after the surgery
  Calculated in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Andjelkov, MD PhD, Principal Investigator — BelPrime Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buschmann J, Gao S, Harter L, Hemmi S, Welti M, Werner CM, Calcagni M, Cinelli P, Wanner GA. Yield and proliferation rate of adipose-derived stromal cells as a function of age, body mass index and harvest site-increasing the yield by use of adherent and supernatant fractions? Cytotherapy. 2013 Sep;15(9):1098-105. doi: 10.1016/j.jcyt.2013.04.009. Epub 2013 Jun 22. PMID 23800730
- [Result] Mojallal A, Lequeux C, Shipkov C, Duclos A, Braye F, Rohrich R, Brown S, Damour O. Influence of age and body mass index on the yield and proliferation capacity of adipose-derived stem cells. Aesthetic Plast Surg. 2011 Dec;35(6):1097-105. doi: 10.1007/s00266-011-9743-7. Epub 2011 May 26. PMID 21614659
- [Result] Faustini M, Bucco M, Chlapanidas T, Lucconi G, Marazzi M, Tosca MC, Gaetani P, Klinger M, Villani S, Ferretti VV, Vigo D, Torre ML. Nonexpanded mesenchymal stem cells for regenerative medicine: yield in stromal vascular fraction from adipose tissues. Tissue Eng Part C Methods. 2010 Dec;16(6):1515-21. doi: 10.1089/ten.TEC.2010.0214. Epub 2010 Sep 6. PMID 20486782